CLINICAL TRIAL: NCT06819215
Title: Phase I/II Clinical Study To Evaluate The Safety, Tolerability, Pharmacokinetics, Pharmacodynamics And Preliminary Efficacy of VB15010 Tablets In Patients With Advanced Solid Tumors
Brief Title: Phase I/II Clinical Study to Evaluate VB15010 Tablets in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Yangli Pharmaceutical Technology Co., Ltd. (Industry)
Collaborators: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB15010-001
Record Dates: First submitted 2025-01-20; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Neoplasms; Neoplasms, Breast; Tumor; PARP; Ovarian Neoplasms; Prostatic Cancer; Pancreatic Cancer; Breast Cancer; Biliary Cancer; Colorectal Cancer
Keywords: VB15010; PARP; Ovarian cancer; Prostatic Cancer; Pancreatic cancer; Breast cancer; Biliary Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): VB15010 Monotherapy
  Interventions: Drug: VB15010

INTERVENTIONS:
Drug: VB15010 — Oral PARP1 inhibitor

SUMMARY:
This research is designed to determine if experimental treatment with PARP1 inhibitor, VB15010 is safe, tolerable, and has anti-cancer activity in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 at the time of screening;
* Histological or cytological confirmation of advanced malignancy ;
* Progressive cancer at the time of study entry;
* Adequate organ and marrow function as defined by the protocol;
* Homologous recombination repair gene mutation.

Exclusion Criteria:

* Major surgery within 4 weeks of the ﬁrst dose of study treatment.
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring continuous corticosteroids at a dose of >10mg prednisone/day or equivalent for at least 4 weeks prior to start of study treatment. Patients with leptomeningeal carcinomatosis are excluded.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with adverse events/serious adverse events | From time of Informed Consent to 30+7 days post last dose
  Number of patients with adverse events and with serious adverse events including abnormal clinical observations, abnormal ECG parameters, abnormal laboratory assessments and abnormal vital signs that changed from baseline
The number of subjects with dose-limiting toxicity (DLT), as deﬁned in the protocol. | At the end of Cycle 1(each cycle is 28 days)
  A DLT is defined as any toxicity that occurs from the ﬁrst dose of study treatment up to and including the planned end of Cycle 1 (the DLT assessment period) that is assessed as unrelated to the disease or disease-related processes under investigation.

SECONDARY OUTCOMES:
Maximum plasma concentration of the drug (Cmax) | At predefined intervals throughout the treatment period (through study completion, an everage of 1 year)
  The concentration of VB15010 in plasma will be determined (Cmax will be derived)
Objective Response Rate (prostate cancer) | From Screening to conﬁrmed progressive disease (approximately 1 year)
  Best response until progression, as deﬁned by RECIST 1.1 or PCWG3 (bone)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Shandong First Medical university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No